CLINICAL TRIAL: NCT06332976
Title: Patients' Preferences for Adjuvant or Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: PrefeRences And ChemoTherapy In Breast Cancer patiEnts
Acronym: PRACTICE
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1521
Record Dates: First submitted 2024-03-18; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Female Breast Cancer
Keywords: Early breast cancer; Locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Before chemotherapy start: Women candidate to adjuvant or neoadjuvant chemotherapy for breast cancer at the time of informed consent (interview before the start of CT)
  Interventions: Other: Completion of questionnaires
- During chemotherapy: Women who are receiving chemotherapy at the time of informed consent (interview within 1 year from beginning of CT)
  Interventions: Other: Completion of questionnaires
- After chemotherapy end: Women who already received chemotherapy at the time of informed consent (interview after more than 4 years of CT end)
  Interventions: Other: Completion of questionnaires

INTERVENTIONS:
Other: Completion of questionnaires — Completion of questionnaires at the time of study entry

SUMMARY:
The aim of the present study is to ask women treated with adjuvant or neoadjuvant chemotherapy for breast cancer what survival benefit would justify the treatment.

The benefit should be evaluated in terms of Survival rate trade off and Survival time trade off value. The analyses will be conducted into three different groups of patients to value the survival benefit expected:

1. before to start the chemotherapy
2. during chemotherapy
3. after the end of chemotherapy

DETAILED DESCRIPTION:
The chemotherapy is generally proposed a large number of early breast cancer patients to reduce the risk of recurrence and death. However chemotherapy is associated with side effects that impact the quality of life of the patients.

Patients are more likely to accept treatment on the basis of presented relative rather than absolute risks and so the question arises as to whether unrealistic improvements in outcome are expected by patients. The interviews with patients in the proposed trial will elicit the expected gains both in terms of survival and life years and will be able to assess the proportion of patients who considered an improvement of realistic size was sufficient to justify the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early or locally advanced breast cancer
* Patients candidate to adjuvant/neoadjuvant chemotherapy or patients who are receiving adjuvant/neoadjuvant chemotherapy or patients who received adjuvant/neoadjuvant chemotherapy
* Sufficient literacy in Italian to complete the questionnaires
* Patients must provide signed, written or advanced electronic signature (AES or AdES), informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients candidate to or who are receiving/have already redceived adjuvant or neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of risk reduction needed to consider adjuvant or neoadjuvant chemotherapy worthwhile | 1 week
  Risk reduction will be evaluated in the 40% and 20% 5 years risk scenarios
Prolonged survival time gain needed to consider CT worthwhile | 1 week
  Prolonged survival time gain will be evaluated in the 5-yr and 15-yr survival scenarios

SECONDARY OUTCOMES:
Behavior assessment | 1 week
  Collection of CONOR questionnaire (minimum value: 0, maximum value: 5 - higher scores mean a greater agreement with the statement)
Reaction to uncertain situations assessment | 1 week
  Collection of Intolerance of Uncertainty Scale Short-Form (IUS-12) questionnaire (minimum value: 1, maximum value: 5 - higher scores mean a greater agreement with the statement)
Regret and disappointment assessment | 1 week
  Collection of Regret and Disappointment Scale (RDS) questionnaire (minimum value: 1, maximum value: 7 - higher scores mean a greater agreement with the statement)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Montagna, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy